CLINICAL TRIAL: NCT02244008
Title: Effects of Anteroposterior Talus Mobilization on Range of Motion, Pain, and Functional Capacity in Participants With Sub-acute and Chronic Ankle Injuries: A Randomized Controlled Trial
Brief Title: Accumulative Effects of Talus Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, RAFAEL DUARTE SILVA, Master, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RDS3123
Record Dates: First submitted 2014-09-15; First posted 2014-09-18 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Ankle Sprains; Ankle Fractures; Ankle Dislocations; Ankle Bruises; Achilles Tendon Rupture
Keywords: Mobilization; Joint Range of Motion; Ankle; Manual Therapy
MeSH Terms: conditions — Ankle Injuries; Ankle Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- joint mobilization (Experimental): Anteroposterior mobilization of the talus (Maitland mobilization grade III)
  Interventions: Other: joint mobilization
- manual contact (Placebo Comparator)
  Interventions: Other: manual contact

INTERVENTIONS:
Other: joint mobilization — The experimental group received joint mobilization (anteroposterior mobilization of the talus - Maitland grade III). During the mobilization cyclic movements were applied in an anteroposterior direction from the first tissue resistance barrier until the end of the accessory range of motion without any pain or discomfort. This mobilization maneuver was performed in 30-second duration sets with a 30-second interval between each set. The interventions lasted two weeks with three sessions each, completing six sessions.
  Arms: joint mobilization
Other: manual contact — The placebo group received only manual contact. This maneuver was performed in 30-second duration sets with a 30-second interval between each set. The interventions lasted two weeks with three sessions each, completing six sessions.
  Arms: manual contact

SUMMARY:
The purpose of this study is to verify the effect of anteroposterior talus mobilization on range of motion, pain, and functional capacity in participants with sub-acute and chronic ankle injuries.

DETAILED DESCRIPTION:
The purpose of this study was to verify the acute effect (one session) and chronic (six sessions) and follow-up of the anteroposterior talus mobilization Maitland's grade III on range of motion, pain, and functional capacity in participants with sub-acute and chronic ankle injuries. Thirty eight volunteers subjects (male and female) participated of this study with minimum 18 and maximum 59 years old. The volunteers were allocated in two groups: experimental and control. The variables related to range of motion, pain and functional capacity were measured by biplane goniometer, Visual Analog Scale and Foot and Ankle Ability Measure respectively in four moments: 1- baseline; 2- after the first intervention; 3- after the sixth intervention (two weeks); 4- follow-up (one month). The experimental group received anteroposterior articular mobilization of the talus and the control group received manual contact.

ELIGIBILITY:
Inclusion Criteria:

* unilateral traumatic injury of the ankle with at least two weeks and maximum eight months
* at least a 5º limitation of passive dorsiflexion in comparison to the contralateral side
* do not be under another physical therapy treatment for the lesion
* able to unload partial or total body weight
* do not be in use of analgesic
* provided informed consent after receiving and explanation of all procedures and pertinent information regarding the study

Exclusion Criteria:

* joint blockage by surgical fixation or ankylosis
* presence of vascular, rheumatic, neurological and neoplastic disease in the lower limb
* open or contagious lesion in the ankle region
* pain during palpation in the region anterior of the ankle

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in dorsiflexion range of motion | 1 month
  Dorsiflexion range of motion were measured by biplane goniometer.

SECONDARY OUTCOMES:
Changes in pain intensity | 1 month
  Pain were measured by Visual Analog Scale.
Changes in functional capacity | 1 month
  Functional capacity were measured by Foot and Ankle Ability Measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Minas Gerais College of Medical Sciences, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Result] Hoch MC, Andreatta RD, Mullineaux DR, English RA, Medina McKeon JM, Mattacola CG, McKeon PO. Two-week joint mobilization intervention improves self-reported function, range of motion, and dynamic balance in those with chronic ankle instability. J Orthop Res. 2012 Nov;30(11):1798-804. doi: 10.1002/jor.22150. Epub 2012 May 18. PMID 22610971
- [Result] Landrum EL, Kelln CB, Parente WR, Ingersoll CD, Hertel J. Immediate Effects of Anterior-to-Posterior Talocrural Joint Mobilization after Prolonged Ankle Immobilization: A Preliminary Study. J Man Manip Ther. 2008;16(2):100-5. doi: 10.1179/106698108790818413. PMID 19119395
- [Result] Teixeira LM, Pires T, Silva RD, de Resende MA. Immediate effect of a single anteroposterior talus mobilization on dorsiflexion range of motion in participants with orthopedic dysfunction of the ankle and foot. J Manipulative Physiol Ther. 2013 Jul-Aug;36(6):369-75. doi: 10.1016/j.jmpt.2013.06.003. Epub 2013 Jul 11. PMID 23850371
- [Result] Hoch MC, McKeon PO. Joint mobilization improves spatiotemporal postural control and range of motion in those with chronic ankle instability. J Orthop Res. 2011 Mar;29(3):326-32. doi: 10.1002/jor.21256. Epub 2010 Sep 30. PMID 20886654
- [Result] Harkey M, McLeod M, Van Scoit A, Terada M, Tevald M, Gribble P, Pietrosimone B. The immediate effects of an anterior-to-posterior talar mobilization on neural excitability, dorsiflexion range of motion, and dynamic balance in patients with chronic ankle instability. J Sport Rehabil. 2014 Nov;23(4):351-9. doi: 10.1123/jsr.2013-0085. Epub 2014 Apr 3. PMID 24700526